CLINICAL TRIAL: NCT03674489
Title: Local and Widespread Hypoalgesic Effects of Neurodynamic Mobilization in Healthy Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brenau University (Other)
Responsible Party: Principal Investigator, Daniel Maddox, PT, DPT, Assistant Professor, Brenau University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1208684-5
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Pain; Pain, Neuropathic
Keywords: neurodynamics; neurodynamic mobilization; quantitative sensory testing; median nerve; pressure pain threshold; thermal pain threshold; thermal pain tolerance
MeSH Terms: conditions — Pain; Neuralgia

STUDY DESIGN:
Intervention Model Description: Each subject will be randomized to one of three groups:
  * Neurodynamic Slider Mobilization
  * Neurodynamic Tensioner Mobilization
  * Sham Neurodynamic Mobilization
  Outcomes will be assessed immediately prior to and immediately following the intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neurodynamic Slider Mobilization (Active Comparator)
  Interventions: Other: Neurodynamic Slider Mobilization
- Neurodynamic Tensioner Mobilization (Active Comparator)
  Interventions: Other: Neurodynamic Tensioner Mobilization
- Sham Neurodynamic Mobilization (Sham Comparator)
  Interventions: Other: Sham Neurodynamic Mobilization

INTERVENTIONS:
Other: Neurodynamic Slider Mobilization — Subjects will be positioned in supine with the examiner supporting his/her arm and facing caudally. The arm will be taken into the ULNT2a position as described in Butler's text - so as to bias the median nerve. Once passive resistance is felt or a feeling of mild tension is reported in the median nerve field, a series of mobilizations will be performed to "slide" the nerve proximally and distally in an alternating manner via providing wrist extension with concurrent shoulder girdle elevation and then providing wrist flexion with concurrent shoulder girdle depression. This will be performed for 2 sets of 10 cycles at a rate of 6 seconds per cycle (3 sec in each position) - not moving further into described tension or passive resistance.
  Other Names: ULNT2a Slider; MNT2 Slider
  Arms: Neurodynamic Slider Mobilization
Other: Neurodynamic Tensioner Mobilization — Subjects will be positioned in supine with the examiner supporting his/her arm and facing caudally. The arm will be taken into the ULND2a position as described in Butler's text - so as to bias the median nerve. Once passive resistance is felt or a feeling of mild tension is reported in the median nerve field, a series of mobilizations will be performed to "tension" the nerve in an alternating on/off manner via providing wrist extension with concurrent shoulder girdle depression and then providing wrist flexion with concurrent shoulder girdle elevation. This will be performed for 2 sets of 10 cycles at a rate of 6 seconds per cycle (3 sec in each position) - not moving further into described tension or passive resistance.
  Other Names: ULNT2a Tensioner; MNT2 Tensioner
  Arms: Neurodynamic Tensioner Mobilization
Other: Sham Neurodynamic Mobilization — Subjects will be positioned in supine with the examiner supporting his/her arm and facing cranially - in a similar position as the UNLD1 test described previously. From here, the therapist will position the patient's arm in 45 deg. of shoulder abduction without scapular depression, 45 deg. of shoulder external rotation, 45 deg. of elbow flexion, and forearm pronation. From this position, a series of sham mobilizations will be performed by passively alternating flexion and extension of the wrist for 2 sets of 10 cycles at a rate of 6 seconds per cycle (3 sec in each position).
  Arms: Sham Neurodynamic Mobilization

SUMMARY:
Background & Significance Pain is the primary reason many patients seek care from healthcare professionals who utilize various manual therapy techniques. Gaining further understanding of the hypoalgesic properties of such techniques can enable practitioners to more skillfully integrate them in managing patients presenting with pain. Previous research has revealed that various manual techniques result in both local and widespread hypoalgesic changes in asymptomatic controls and patients in pain. Much of this previous research has investigated thrust manipulation; however, there is a paucity of similar research investigating these effects in neurodynamic mobilization.

Specific Aims Aim: To assess for immediate local and widespread hypoalgesic effects of neurodynamic mobilization applied to the upper extremity.

Hypotheses:

* Subjects who receive neurodynamic mobilizations will exhibit greater positive changes in local and widespread Qualitative Sensory Testing (QST) measures compared to those who receive a sham mobilization.
* Subjects who receive neurodynamic mobilizations will exhibit greater positive changes in elbow ROM and reported sensation intensity with upper limb neurodyndamic testing as compared to those who receive a sham mobilization.

Aim: To assess for differences in immediate local and widespread hypoalgesic effects of sliding vs tensioning neurodynamic mobilization techniques applied to the upper extremity

Hypotheses:

* Subjects who receive sliding neurodynamic mobilizations will exhibit greater positive changes in local and widespread QST measures compared to those who receive tensioning neurodynamic mobilization
* Subjects who receive sliding neurodynamic mobilizations will exhibit greater positive changes in elbow range of motion (ROM) and reported sensation intensity with upper limb neurodynamic testing testing compared to those who receive a tensioning neurodynamic mobilization

DETAILED DESCRIPTION:
See protocol uploaded in documents section

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65
* Ability to speak and comprehend English.

Exclusion Criteria:

* Current neck or upper extremity symptoms
* Disorders that could result in impaired sensation - such as diabetes.
* Current use of prescription pain medication or other medications that could result in altered pain perception - such as anti-anxiety medications or anti-depressants.
* History of any chronic painful condition
* Diagnosis of any major psychiatric disorder
* Current pregnancy
* Any painful condition within the past 3 months for which care was sought

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) | change from baseline immediately after intervention
  PPT will be assessed bilaterally over the thenar eminences, over the dorsal aspect of the 1st carpometacarpal (CMC) joint, and over the tibialis anterior using a pressure algometer with an affixed 1cm2 rubber tip.
Thermal Pain Threshold (TPT) | change from baseline immediately after intervention
  TPT will be assessed bilaterally over the thenar eminences, over the dorsal aspect of the 1st carpometacarpal (CMC) joint, and over the tibialis anterior.
Thermal Pain Tolerance (TPTol) | change from baseline immediately after intervention
  TPTol will be assessed bilaterally over the thenar eminences, over the dorsal aspect of the 1st carpometacarpal (CMC) joint, and over the tibialis anterior.
Elbow Extension ROM Obtained on Neurodynamic Testing | change from baseline immediately after intervention
  A neurodynamic test of the median nerve will be performed according to the ULNT1 procedure originally described by David Butler. Degrees of elbow extension will then be recorded using a universal goniometer, and each subject will rate each of the following 5 sensory descriptors on a 10 cm Visual Analog Scale (VAS): "Stinging", "Tingling", "Tightness", "Sharpness", and "Numbness". The average of the 5 sensory descriptor ratings will then be averaged to create a single sensory descriptor VAS score - as outlined in Beneciuk et al 2009.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Maddox, DPT, Principal Investigator — Brenau University
Locations (1):
- Brenau University, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No